CLINICAL TRIAL: NCT07198178
Title: The Effect of Peer Support on The Clinical Readiness of First Year Nursing Students
Acronym: Peer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senem Duman (Other)
Responsible Party: Sponsor-Investigator, Senem Duman, Lecturer, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SaglikBilimleriU-2
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: First Year Students
Keywords: nursing student; peer support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): First-year nursing students participated in the clinical practice and agreed to participate in the study. Data collection forms were applied before, during, and after the clinical practice. No intervention was performed.
- Intervention group (Experimental): The participants were first-year nursing students who agreed to participate in the study. These students were enrolled in a peer support program. Data collection forms were administered before, during, and after clinical practice.
  Interventions: Other: Peer Training

INTERVENTIONS:
Other: Peer Training — Peer Selection Fourth-year nursing students who have completed the Clinical Practice-I course and are currently attending the Clinical Practice-II course and are in clinical practice four days a week will be invited to volunteer to become peer tutors after being informed about the purpose of the study. These volunteer peer tutors will be selected from among students with strong academic achievement (grade point average of 3.50 or above) and good communication skills, taking into account their clinical experience.
  Peer Training Fourth-year students selected as peers will receive a training program consisting of four 40-minute sections, each lasting 160 minutes, prepared by the faculty members and aligned with the Fundamentals of Nursing course curriculum. This training aims to equip peers with the knowledge and skills to guide, provide feedback, and support to first-year students during clinical practice. The training will utilize active learning methods such as role-playing and case st
  Arms: Intervention group

SUMMARY:
Nursing students' first clinical practice experiences are one of the most anxiety-inducing and stressful aspects of nursing education. Nursing students experience anxiety due to fear of making mistakes in clinical practice, clinical practice grades, reactions from patients and their relatives, reactions from clinic staff, and a lack of theoretical knowledge. This anxiety can hinder learning and work habits, reduce motivation, and negatively impact skill development and clinical readiness. To prevent or minimize these negative effects, faculty members should take precautions and develop supportive alternative educational methods in addition to traditional educational approaches. Supporting nursing students with peer tutoring is known to have positive effects on clinical readiness. A study on anxiety and clinical performance among nursing students found that they experienced anxiety during clinical practice. Another study found that students who received skills training through a peer tutoring model learned skills more easily and retained them. The peer support nursing students received during clinical practice increased their sense of security, increased their motivation, and facilitated a more rapid improvement in their clinical readiness. The purpose of this study was to examine the effects of peer education received by first-year nursing students during their first clinical practice on clinical readiness and stress levels. This study emphasizes the importance of peer support in nursing education programs. It is expected that peer support provided to first-year nursing students using the peer education model will reduce the anxiety students experience during their first clinical practice and positively contribute to their clinical readiness.

The research population consisted of 20 first-year students in the Department of Nursing at a state university. The sample size of the study was determined through power analysis using the G-Power 3.1.9.7 program. A two-sided hypothesis test with 95% confidence, 95% test power (α=0.05, 1-β=0.95), and an effect size of d=0.8 was used to test the study. A minimum sample size of 84 students, with at least 42 in each group, was determined for a total of 92 students. Considering the possibility of data loss due to withdrawal requests and absenteeism during the study, an additional 10% of the calculation was taken to include 92 students (Experimental: 46, Control: 46). The study included first-year students in the Faculty of Nursing during the 2024-2025 academic year, who had no vision or hearing impairments, were participating in clinical practice for the first time, had no first-degree family members who were healthcare professionals, and volunteers.

Intervention Peer Selection Fourth-year nursing students who have completed the Clinical Practice-I course and are attending the Clinical Practice-II course and are practicing clinically four days a week will be informed about the purpose of the study and invited to volunteer to be peer educators. These volunteer peer educators will be selected from among students with strong academic achievement (grade point averages of 3.50 and above) and good communication skills, taking into account their clinical experience.

Peer Training Fourth-year students selected as peers will receive a training program consisting of four 40-minute sections, each lasting 160 minutes, tailored to the Fundamentals of Nursing course curriculum and prepared by the faculty. This training aims to equip peers with the knowledge and skills to guide, provide feedback, and support to first-year students during clinical practice. The training will utilize active learning methods such as role-playing and case studies.

Peer Support Implementation Process Peer support aims to help first-year students and those experiencing their first clinical practice experience feel more confident, increase their motivation, and develop their clinical skills. Peer support sessions will be delivered one-on-one in a hospital setting during the Fundamentals of Nursing course. Each first-year student will be paired with a fourth-year peer. Peer support will be actively implemented throughout the 10-day clinical practice period.

Data Collection Tools Introductory Information Form Perceived Stress Scale for Nursing Students (Pretest-Posttest) Clinical Practice Readiness Scale for Nursing Students (Pretest-Posttest) Peer Mentoring Rating Scale (Posttest) Research Hypotheses H1: Peer support has an effect on the clinical readiness levels of first-year nursing students.

H2: Peer support has an effect on the stress levels of first-year nursing students.

H3: Peer support has an effect on the clinical practice anxiety levels of first-year nursing students.

ELIGIBILITY:
Inclusion Criteria:

* The study will include first-year students at the Faculty of Nursing in the 2024-2025 academic year, students who do not have vision or hearing problems, students who are involved in clinical practice for the first time, students whose first-degree family members are not healthcare professionals, and volunteers.

Exclusion Criteria:

* Not meeting the criteria for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
At the Beginning of Work | Baseline (Just before peer pairing)
  Before Clinical Practice, data collection forms were applied to all students who accepted the study.

SECONDARY OUTCOMES:
First Day of Clinical Practice | First 1 day of clinical practice
  Before Clinical Practice, data collection forms were applied to all students who accepted the study.

OTHER OUTCOMES:
After Clinical Application | Last 1 day of clinical practice
  After Clinical Practice, both mentors and mentees applied data collection forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No